CLINICAL TRIAL: NCT06294327
Title: Comparing a REactive STatic Air Mattress to an Alternating Air Pressure Mattress in the Prevention of Pressure Ulcers: a Randomized Controlled Trial (RESTART)
Brief Title: RESTART the Prevention of Pressure Ulcers: Comparing the Effectiveness and Cost of a Reactive Static Air Mattress and Alternating Air Pressure Mattress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaz (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC23027
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Pressure Injury; Pressure Ulcer; Decubitus Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reactive static air support surfaces (Repose®) (Experimental): Intervention with Repose® devices
  Standard repositioning protocol is applied.
  Interventions: Device: Reactive static air support surfaces
- Alternating air pressure mattress (ArjoHuntleigh® Alpha Response) (No Intervention): Standard care with mattress type: ArjoHuntleigh® Alpha Response
  Standard repositioning protocol is applied.

INTERVENTIONS:
Device: Reactive static air support surfaces — * Repose® Mattress
  * Repose® Cushion
  * Repose® Wedge
  * Repose® Foot Protectors
  Other Names: Repose® devices
  Arms: Reactive static air support surfaces (Repose®)

SUMMARY:
Pressure ulcers are a global issue and substantial concern for healthcare systems. A review of the literature between January 2000 and December 2012 has revealed that prevalence rate of pressure ulcers in aged care facilities were between 4.1% and 32.2%, and the incidence rates ranged from 1.9% to 59%. Similarly, a systematic review reported that the prevalence of pressure ulcer varied between 0.3% and 46%, and the incidence of pressure ulcer ranged from 0.8% to 34%. Most epidemiological data were obtained from hospitals (38.7%) and institutional long-term care facilities (29.7%).

The costs associated with pressure ulcers are considerable. According to the Agency for Healthcare Research & Quality (2011), the US healthcare system has allocated approximately $ 9.1 - $ 11.6 billion annually for the health care cost of pressure ulcer. In addition to direct treatment-related costs, the development of pressure ulcer also results in litigation and government penalties, and affects hospital performance metrics. A systematic review has reported that the cost for treatment of pressure ulcer was higher than its prevention. That is, the cost per patient per day ranged from € 1.71 to € 470.49 (for treatment) and from € 2.65 to € 87.57 (for prevention) across all settings.

This randomized controlled trial will be performed in a general hospital in a random sample of 308 patients (nursing wards geriatric n=3 and orthopedic (n=3)) who are at high risk of developing pressure ulcers. Patients will be included in the study for a period > 2 hospitalisation days. Skin assessment and risk factor registration will be done on a daily base by the ward nurses. Reliability checks and time measurements will be completed by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Norton score < 14
* Bed and/or chairfast
* no pressure ulcers or at least pressure ulcer category I

Exclusion Criteria:

* Norton Score >/=14
* Pressure ulcers category II, III, IV, deep tissue injury (DTI) or unstageable pressure ulcer
* Expected length of hospital stay < 2 days
* Medical contraindication for use of reactive static air support surfaces
* End of life care (or Do Not Reanimate (DNR) code IV)
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pressure ulcer, category > I | After admission
  Development of a pressure ulcer category > I

SECONDARY OUTCOMES:
Cost of alternating air pressure mattress compared to reactive static air support surfaces | After admission
  Economic cost (€)
Patient comfort | After admission
  To measure the degree of comfort a five point Likert scale was used (1 - 'not comfortable at all', 2 - 'not very comfortable', 3 - 'more or less comfortable', 4 - 'very comfortable', and 5 - 'totally comfortable')

CONTACTS AND LOCATIONS:
Locations (1):
- Vitaz (General Hospital), Sint-Niklaas, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anrys C, Van Tiggelen H, Verhaeghe S, Van Hecke A, Beeckman D. Independent risk factors for pressure ulcer development in a high-risk nursing home population receiving evidence-based pressure ulcer prevention: Results from a study in 26 nursing homes in Belgium. Int Wound J. 2019 Apr;16(2):325-333. doi: 10.1111/iwj.13032. Epub 2018 Nov 9. PMID 30412652
- [Background] Shi C, Dumville JC, Cullum N, Rhodes S, Leung V, McInnes E. Reactive air surfaces for preventing pressure ulcers. Cochrane Database Syst Rev. 2021 May 7;5(5):CD013622. doi: 10.1002/14651858.CD013622.pub2. PMID 33999463
- [Background] Beeckman D, Serraes B, Anrys C, Van Tiggelen H, Van Hecke A, Verhaeghe S. A multicentre prospective randomised controlled clinical trial comparing the effectiveness and cost of a static air mattress and alternating air pressure mattress to prevent pressure ulcers in nursing home residents. Int J Nurs Stud. 2019 Sep;97:105-113. doi: 10.1016/j.ijnurstu.2019.05.015. Epub 2019 Jun 8. PMID 31234104
- [Background] Serraes B, van Leen M, Schols J, Van Hecke A, Verhaeghe S, Beeckman D. Prevention of pressure ulcers with a static air support surface: A systematic review. Int Wound J. 2018 Jun;15(3):333-343. doi: 10.1111/iwj.12870. Epub 2018 Mar 5. PMID 29504266
- See also: SKIN INTEGRITY RESEARCH GROUP (SKINT) — https://www.skintghent.be/en
- See also: University — https://www.ucvvgent.be/
- See also: Study location; VITAZ (general) Hospital and Health Care VITAZ, Moerlandstraat 1, B-9100 Sint-Niklaas Belgium — https://vitaz.be/